CLINICAL TRIAL: NCT06271317
Title: Evaluation of Possible Postoperative Complications After Nissen Sleeve Gastrectomy. French Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_CL_001
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: Nissen sleeve gastrectomy; Morbidity-Fistula-Bariatric surgery; Sleeve gastrectomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nissen sleeve gastrectomy: Nissen sleeve gastrectomy patients
- Sleeve gastrectomy with the data of PMSI: Sleeve gastrectomy with the data of PMSI

SUMMARY:
The purpose of this study is to evaluate the impact about complications between the procedure (sleeve gastrectomy technique with a Nissen fundoplication (N-Sleeve)) and conventional sleeve gastrectomy technique

DETAILED DESCRIPTION:
Obesity is currently a major health problem. 2% of the French adult population is morbidly obese (BMI>40kg/m²). In this case, the only effective treatment is bariatric surgery. More than 50,000 acts of bariatric surgery were performed in 2018 in France. Three main operations are considered: Sleeve Gastrectomy (SG), Roux en Y Gastric Bypass (RYGB) and Gastric Banding.

SG was validated by the Haute Autorité de Santé (HAS) in 2008 and is the most widely used procedure in France (35,580 operations in 2018). It consists of a 2/3 partial gastrectomy. Long-term weight loss of 61 ± 23% is expected, with significant improvement in obesity-related comorbidities.

However, this technique is associated with postoperative complications. Gastric fistula (2%), most often located at the upper end of the stapling line, bleeding from the gastric section (2%) and gastric stenosis (1%) are the most frequent early postoperative complications that may require reoperation. In addition, gastroesophageal reflux disease (GERD) is very common (30-57%), and can have serious consequences for the esophageal mucosa (esophagitis, Barrett's esophagus, cancer). Alarmingly high rates of Barrett's esophagus (17-18%) after SG have recently been described in the long term, causing concern in the medical community. This may be an exacerbation of preoperative GERD symptoms or "de novo" postoperative GERD. Medical treatment is generally effective (proton pump inhibitors (PPIs)). However, the long-term safety of PPIs has not been demonstrated. What's more, these patients' quality of life may be considerably reduced, and re-intervention (gastric Y-bypass) may be necessary to treat refractory GERD.

The classic surgical treatment for GERD, independently of bariatric surgery, is fundoplication, which can be partial (180°: Toupet technique) or total (360°: Nissen technique). The gastric fundus is wrapped around the esophagus to reinforce the esophageal sphincter.

Nissen-Sleeve Gastrectomy (Nissen-SG) is an innovative technique performed in expert centers in France. It consists in creating a total anti-reflux fundoplicature (Nissen) before performing a SG.

A prospective non-comparative pilot study of 25 patients who underwent Nissen-SG in 2014 at Montpellier University Hospital, showed that while 92% of patients had symptoms of GERD preoperatively, 24% were symptomatic at 3 months after Nissen and SG, only 12% had clinical GERD at 6 months and 1 year postoperatively. Excess weight loss at 1 year was 59%, similar to the efficacy of conventional SG, although a larger gastric residual volume was left after Nissen-SG but used as plication. The 5-year results were presented at the SOFFCO 2020 congress and at the International Federation of Obesity Surgery (IFSO) congress. Excess weight loss (EWL) was 70.87% (112 patients) and 58.32% (31 patients) at 2 and 5 years follow-up. Less than 7% of patients had GERD symptoms at 5 years.

Our hypothesis is that the creation of a total anti-reflux fundoplicature prior to performing SLEEVE could significantly reduce the rate of postoperative GERD observed with standard SLEEVE.

What's more, the creation of a Nissen fundoplicature means that a gastric section is made away from the HIS angle (the area most at risk of fistula (90%)), which could reduce this complication almost definitively (no gastric fistula on the staple line in this pilot study).

Quality of life and socio-economic impact could be significant if such hypotheses are confirmed. However, complications specific to the Nissen sleeve, such as dilatation and perforation of the envelope, were also reported in this prospective trial. A 3.9% rate of perioperative complications after Nissen Sleeve was described after the learning curve of the procedure on 301 patients (2018-2020).

Our aim in this study is to highlight that there are no more complications when performing Nissen-SG than SG (taking published PMSI data) and to show a decrease in post-operative GERD after Nissen-SG. To achieve this, data will be collected on patients undergoing Nissen-SG surgery in 2022 until 2024 in 18 French hospitals. For these patients, any post-operative complications and the presence/evolution of GERD will be collected and compared with SG data available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures
* Subjects must be covered by public health insurance
* Contraception efficacy
* Subjects eligible for sleeve gastrectomy after multidisciplinary evaluation according to HAS 2009 criteria: BMI ≥ 40 kg / m² with failure of the dietary treatment for at least 1 year, or a BMI ≥ 35kg / m² with at least one co-morbidity that could be improved after surgery (hypertension, obstructive sleep apnea hypopnea syndrome (OSAHS) and other severe respiratory disorders, severe metabolic disorders (especially type 2 diabetes), debilitating musculoskeletal diseases, non-alcoholic steato-hepatitis (NASH))

Exclusion Criteria:

* Subject unable to read or/and write
* Planned longer stay outside the region that prevents compliance with the visit plan
* Current pregnancy
* Previous bariatric surgery (ring, vertical banded gastroplasty, sleeve gastrectomy or Gastric Bypass).
* Previous reflux surgery
* BMI > 50 kg / m² for women and > 45kg / m² for men (dissecting the hiatus region can be a technical challenge in these cases).
* Barrett oesophagus and esophagitis stage III and IV.
* Funditis
* No affiliation at the French social security scheme.
* Major protected by law.
* Deprivation of liberty by judicial or administrative decision. Participation to another clinical research program.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for sleeve gastrectomy after multidisciplinary evaluation according to HAS 2009 criteria: BMI ≥ 40 kg / m² with failure of the dietary treatment for at least 1 year, or a BMI ≥ 35kg / m² with at least one co-morbidity that could be improved after surgery (hypertension, obstructive sleep apnea hypopnea syndrome (OSAHS) and other severe respiratory disorders, severe metabolic disorders (especially type 2 diabetes), debilitating musculoskeletal diseases, non-alcoholic steato-hepatitis (NASH))
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Study postoperative morbidity after nissen sleeve gastrectomy in Nantes | 30 days post operation
  Collection of complications at 30 days post-op (aphagia, valve necrosis, fistula, etc.) and classification according to Dindo-Clavien.
postoperative morbidity of nissen sleeve gastrectomy with sleeve gastrectomy in France | 30 days post operation
  Comparison of Nissen Sleeve Gastrectomy data at 30d post-op (aphagia, valve necrosis, fistula...) with published PMSI sleeve gastrectomy data.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France